CLINICAL TRIAL: NCT02372240
Title: VLX1570 and Low-Dose Dexamethasone in Relapsed or Relapsed and Refractory Multiple Myeloma: A Clinical and Correlative Phase 1/2 Study
Brief Title: A Study of VLX1570 and Dexamethasone in Myeloma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Dose limiting tox is observed. Study put on full clinical hold.
Sponsor: Vivolux AB (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V14-11056
Record Dates: First submitted 2015-02-05; First posted 2015-02-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — VLX1570; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VLX1570 and dexamethasone (Experimental): VLX1570 IV (0.05, 0.15, 0.3, 0.6, 1.2, 2.0 mg/kg) on days 1, 2, 8, 9, 15 and 16 of a 28-day cycle
  Dexamethasone 20 mg PO/IV
  Interventions: Drug: VLX1570 and dexamethasone

INTERVENTIONS:
Drug: VLX1570 and dexamethasone

SUMMARY:
This is a phase 1/2 single arm study to determine the safety and efficacy of VLX1570 IV infusion administered with low dose dexamethasone in patients with relapsed or relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a phase 1/2, open label study to determine the safety and efficacy of VLX1570 intravenous (IV) infusion administered with low dose dexamethasone on days 1, 2, 8, 9, 15, 16 of a 28-day cycle in patients with confirmed diagnosis of multiple myeloma with relapsed or relapsed and refractory disease (RRMM).

The phase 1 trial design follows an Initial Accelerated Titration design followed by a traditional "3+3" cohort design to establish maximum tolerated dose (MTD) and recommended phase 2 dose (RPTD) for the phase 2 portion of the study. It is anticipated that patients will receive 6 treatment cycles. In the absence of unacceptable toxicity and disease progression, patients have the option of continuing treatment beyond 6 cycles, if the investigator determines that the patient may benefit further from it.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed or relapsed and refractory multiple myeloma following at least 2 prior therapies which must include at least one immunomodulatory drug (e.g., thalidomide, lenalidomide or pomalidomide) and one proteasome inhibitor (e.g., bortezomib or carfilzomib). Patients must not be candidates for regimens known to provide clinical benefit.
2. Measurable disease defined by 1 or more of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL
   * Urine monoclonal protein >200 mg/24 hour
   * Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio (reference 0.26-1.65)
3. Estimated glomerular filtration rate (GFR) ≥30 mL/min as assessed by CKD-epi, MDRD or the Cockcroft-Gault Equation
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
6. Females of child-bearing potential* must have a negative pregnancy test.
7. Males and females of child-bearing potential*, willing to use an effective form of contraception during chemotherapy treatment and for at least 6 months thereafter. Such methods include: (if using hormonal contraception this method must be supplemented with a barrier method, preferably male condom)

   * oral, intra-vaginal or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition for ovulation
   * oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation.
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomised partner
   * true sexual abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of the trial, and withdrawal are not acceptable methods of contraception.
8. Absolute neutrophil count (ANC) ≥1.0 x 109 /L, hemoglobin ≥8 g/dL, and platelet count ≥ 75 x 109/L.
9. Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 2.5 x ULN.
10. Patient has or is willing to have a central venous catheter (e.g. PICC, Port-A-Cath®, Hickman® catheter) for drug administration.

Exclusion Criteria:

1. Any concurrent treatment that would compromise the study including but not limited to:

   * Planned concurrent treatment for multiple myeloma other than bisphosphonates
   * Ongoing corticosteroids for indications other than multiple myeloma allowed as long as the dose does not exceed 10 mg of prednisone per day or equivalent
   * Persisting effects of any previous or ongoing treatment ≥ grade 1 that might compromise delivery of study treatment or assessment of adverse events (except alopecia or neuropathy ≤ grade 2 without pain)
2. Any cytotoxic or biologic therapy less than 2 weeks prior to initiation of therapy.
3. Pregnant or breast feeding females.
4. Uncontrolled hypertension or diabetes.
5. Known active hepatitis B or C infection or HIV infection.
6. Significant cardiovascular disease with NYHA Class III or IV symptoms, or hypertrophic cardiomegaly, or restrictive cardiomegaly, or myocardial infarction within 6 months prior to enrollment, or unstable angina, or unstable arrhythmia.
7. QTc interval >460 msec (males) or >470 msec (females); or repeated demonstration of a QTc interval >450 msec.
8. A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
9. The use of concomitant medications that prolong the QT/QTc interval.
10. Uncontrolled intercurrent illness including but not limited to psychiatric illness/social situations that, in the opinion of the Investigator, would compromise compliance of study requirements or put the patient at unacceptable risk.
11. Active infection requiring systemic treatment within one week prior to first dose.
12. Major surgery within 1 month prior to enrollment.
13. Use of any investigational agent within the last 28 days. For classes of investigational agents that are not known to have prolonged toxicities the wash-out time may be decreased to 14 days after agreement with the Medical Monitor.
14. History of other malignancy (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma) except if the patient has been free of symptoms and without active therapy for at least 2 years.
15. Known intolerance to steroids or H1/H2-antagonists.
16. Serum calcium (corrected for albumin) level above the ULN range (treatment of hypercalcemia is allowed and subject may enroll if hypercalcemia returns to normal with standard treatment).
17. Diagnosed with plasma cell leukemia, POEMS syndrome or amyloidosis.
18. Patients with a history of ventral nervous system (CNS) myeloma or other CNS malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of VLX1570 with low dose dexamethasone | Duration of treatment (expected avg. 6 months) and up to 30 days following the last dose/off-study
Clinical benefit rate (minimal response or better) in patients associated with administration of VLX1570 with low dose dexamethasone | From date of first dose until the date of first documented progression or date of death from any cause, whichever comes first, up to 2 years

SECONDARY OUTCOMES:
Frequency and severity of adverse events associated with the combination of VLX1570 and low dose dexamethasone | Duration of treatment (expected avg. 6 months) and up to 30 days following the last dose/off-study
Pharmacokinetic profile of VLX1570 following IV infusion | 48 hours post dose
  PK parameters include Cmax, Tmax, AUC, half-life, clearance
Investigate Objective Response per International Myeloma Working Group criteria at any dose of VLX1570 with low dose dexamethasone. | Pre-dose cycle 1, 2 and cycles on new dose, and in cycle 5 (or at time of CR or PD).
  SPEP/UPEP, IFE, SFLC

OTHER OUTCOMES:
Blood, bone marrow and other tissues collected during study, will be used for biomarker and mechanism of action studies | Pre-dose each day 16 of each new cycle on new dose and in cycle 5 (or at time of CR or PD)
  May include examination of gene expression, proteomics and functional analysis or proteasomes, proteasomal subunits and associated enzymes

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States